CLINICAL TRIAL: NCT02906865
Title: Proximal Hamstring Avulsion Surgery Cohort Study
Acronym: PHAS
Status: Recruiting | Type: Observational
Sponsor: Fonds de Dotation pour la Recherche Clinique en Orthopédie et Pathologie du Sport (Other)
Responsible Party: Sponsor
Other Study IDs: PHAS
Record Dates: First submitted 2016-09-13; First posted 2016-09-20 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Proximal Hamstring Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Proximal hamstring tendons repair — Proximal hamstring tendons repair

SUMMARY:
Proximal hamstring rupture is a rare injury, which may be immediately diagnosed.

In 1996, Sallay showed that functional results of surgical repair were better than those of conservative treatment. Surgery is now the rule. The main aim of this study is to obtain a more detailed and quantified description of the postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* a partial or complete hamstring proximal rupture,
* treated surgically
* diagnosis of rupture based on clinical signs and confirmed on MRI

Exclusion Criteria:

* no exclusion criteria

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Partial or complete hamstring proximal rupture
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2002-01; Primary Completion 2020-01 (Actual); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Activity level | 2 years
  UCLA (University of California, Los Angeles ) score

SECONDARY OUTCOMES:
Return to sports | 1 year
  Yes/no
Healing on MRI | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique du Sport, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lefevre N, Bohu Y, Naouri JF, Klouche S, Herman S. Returning to sports after surgical repair of acute proximal hamstring ruptures. Knee Surg Sports Traumatol Arthrosc. 2013 Mar;21(3):534-9. doi: 10.1007/s00167-012-2204-2. Epub 2012 Sep 13. PMID 22972314
- [Result] Lefevre N, Bohu Y, Klouche S, Herman S. Surgical technique for repair of acute proximal hamstring tears. Orthop Traumatol Surg Res. 2013 Apr;99(2):235-40. doi: 10.1016/j.otsr.2012.05.006. Epub 2012 Aug 25. PMID 22926295
- [Derived] Lefevre N, Moussa MK, El Otmani L, Valentin E, Meyer A, Grimaud O, Bohu Y, Hardy A. Surgical Treatment of Proximal Hamstring Avulsion Injuries Compared With Nonsurgical Treatment: A Matched Comparative Study With a Mean Follow-up of >4 Years From the Proximal Hamstring Avulsion Surgery Cohort Study. Am J Sports Med. 2024 Sep;52(11):2718-2727. doi: 10.1177/03635465241270139. Epub 2024 Aug 21. PMID 39165177
- [Derived] Lefevre N, Moussa MK, Valentin E, Meyer A, Bohu Y, Gerometta A, Khiami F, Grimaud O, Khalaf Z, Hardy A. Predictors of Early Return to Sport After Surgical Repair of Proximal Hamstring Complex Injuries in Professional Athletes: A Prospective Study. Am J Sports Med. 2024 Mar;52(4):1005-1013. doi: 10.1177/03635465231225486. Epub 2024 Feb 14. PMID 38353018